CLINICAL TRIAL: NCT00456183
Title: A Phase I Study Evaluating the Safety and Immunogenicity of a New TB Vaccine, MVA85A, in Healthy Volunteers Who Are Latently Infected With Mycobacterium Tuberculosis.
Brief Title: Safety and Immunogenicity of MVA85A in Volunteers Latently Infected With TB.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB007
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-05-31 (Estimated); Status verified 2007-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Latent; TB; Vaccine; MVA 85A
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MVA 85A

SUMMARY:
This study is designed to evaluate the safety of MVA85A in healthy volunteers in the UK who are latently infected with M.tb. A single vaccination with MVA85A, when administeredat a dose of 5 x 107pfu intradermally, is safe in both mycobacterially naïve individuals and those previously vaccinated with BCG. We will use the same vaccination regime in this study. Subjects will be defined as being latently infected if they have a positive elispot response to ESAT6 or CFP10. Subjects will be identified from TB contact clinics.

DETAILED DESCRIPTION:
Tuberculosis (TB) kills about three million people annually. It is estimated that one third of the world's population are latently infected with Mycobacterium tuberculosis (M.tb) (Dye, 1999). These latently infected individuals are at risk of reactivation of infection, should they become immunosuppressed. Worldwide, coinfection with HIV is the commonest cause of immunosuppression and increases the chances of reactivation from a 10% lifetime risk to a 10% annual risk (Corbett, 1996). The currently available vaccine, M. bovis BCG, is largely ineffective at protecting against adult pulmonary disease in endemic areas and it is widely agreed that a new more effective tuberculosis vaccine is a major global public health priority (Colditz, 1994). However, it may be unethical and impractical to test and deploy a vaccine strategy that does not include BCG, as BCG does confer worthwhile protection against TB meningitis and leprosy. An immunisation strategy that includes BCG is also attractive because the populations in which this vaccine candidate will need to be tested will already have been immunised with BCG. Given the high prevalence of infection with M.tb, a vaccine that could be administered to latently infected individuals and eradicate latent infection would have an enormous impact on the mortality and morbidity from TB.

M.tb is an intracellular organism. CD4+ Th1-type cellular responses are essential for protection and there is increasing evidence from animal and human studies that CD8+ T cells also play a protective role (Flynn, 2001). However, it has generally been difficult to induce strong cellular immune responses in humans using subunit vaccines. DNA vaccines, recombinant viral vectors and protein/adjuvant combinations all induce both CD4+ and CD8+ T cells, however none of these antigen delivery systems induce high levels of antigen specific T cells, when used alone. Heterologous prime-boost immunisation strategies involves giving two different vaccines, each encoding the same antigen, several weeks apart. Using a DNA prime-recombinant modified vaccinia virus Ankara (MVA) boost induces higher levels of antigen specific CD4+ and CD8+ T cells than using homologous boosting with the same vector in a number of different disease models (Schneider, 1998; McShane, 2001). Given the protective efficacy of BCG in childhood, ideally BCG would be the priming immunisation in such a prime-boost strategy. In order to do this, we have focused on antigen 85A as a candidate antigen.

Antigen 85A is highly conserved amongst all mycobacterial species and is present in all strains of BCG. Antigen 85A is a major secreted antigen from M. tuberculosis which forms part of the antigen 85 complex (A, B and C). This complex constitutes a major portion of the secreted proteins of both M.tb and BCG. It is involved in fibronectin binding within the cell wall and has mycolyltransferase activity. Antigen 85A is immunodominant in murine and human studies and is protective in small animals (Huygen, 1996). Recombinant modified vaccinia virus Ankara (rMVA). Many viruses have been investigated as potential recombinant vaccines. The successful worldwide eradication of smallpox via vaccination with live vaccinia virus highlighted vaccinia as a candidate for recombinant use. The recognition in recent years that nonreplicating strains of poxvirus such as MVA and avipox vectors can be more immunogenic than traditional replicating vaccinia strains has enhanced the attractiveness of this approach. MVA (modified vaccinia virus Ankara) is a strain of vaccinia virus which has been passaged more than 570 times though avian cells, is replication incompetent in human cell lines and has a good safety record. It has been administered to more than 120,000 vaccinees as part of the smallpox eradication programme, with no adverse effects, despite the deliberate vaccination of high risk groups (Stickl, 1974; Mahnel, 1994). This safety in man is consistent with the avirulence of MVA in animal models. MVA has six major genomic deletions compared to the parental genome severely compromising its ability to replicate in mammalian cells (Meher, 1991). No replication has been documented in nontransformed mammalian cells. Viral replication is blocked late during infection of cells but importantly viral and recombinant protein synthesis is unimpaired even during this abortive infection. The viral genome has been proven to be stable through a large series of passages in chicken embryo fibroblasts. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. When tested in animal model studies recombinant MVAs have been shown to be avirulent, yet protectively immunogenic as vaccines against viral diseases and cancer. Recent studies in severely immuno-suppressed macaques have supported the view that MVA should be safe in immuno-compromised humans (Akira, 2001; Stittelaar, 2001). There is now safety data from a number of recombinant MVAs that are currently in Phase I/II trials in both the UK and Africa. Useful data on the safety and efficacy of various doses of a recombinant MVA vaccine comes from clinical trial data with a recombinant MVA expressing a number of CTL epitopes from Plasmodium falciparum pre-erythrocytic antigens fused to a complete pre-erythrocytic stage antigen, Thrombospondin Related Adhesion Protein (TRAP). To date MVA ME-TRAP has been administered to over 250 healthy volunteers in Oxford and The Gambia without any serious adverse events (Adrian Hill, personal communication). Volunteers have received one to three doses of from 3 to 15 x 107 pfu per dose of intra-dermal vaccine at three-week intervals. All subjects have temporary local redness with typically a 5mm central red area with a paler pink surrounding area that ranges in size from about 1 -7cm in diameter and peaks at 48 hours post vaccination. At seven days post vaccination generally only the central red area remains. This fades over the next few weeks and is usually not apparent at 2 months after vaccination. The emerging safety profile of recombinant MVA vaccine is supported by data from clinical studies of three other MVA recombinants made in Oxford and currently in clinical studies using MVAs for HIV, HBV and melanoma. Recombinant MVA encoding antigen 85A MVA85A induces both a CD4+ and a CD8+ epitope when used to immunise mice. When mice are primed with BCG and then given MVA85A as a boost, the levels of CD4+ and CD8+ T cells induced are higher than with either BCG or MVA85A alone, and this regime is more protective than either vaccine alone (Goonetilleke et al, 2003). In the more sensitive guinea pig model, guinea pigs vaccinated with BCG, and then MVA85A, and then a second viral vector, fowlpox expressing antigen 85A, 6/6 guinea pigs are alive at the end of the experiment, compared with 2/6 guinea pigs vaccinated with BCG alone, and 0/6 control animals (Williams et al, submitted). In rhesus macaques, this BCG prime-MVA85A and Fowlpox85A boost is more immunogenic than any of the vaccines alone. Clinical studies using MVA85A MVA85A (at a dose of 5 x 107pfu) has been administered to 40 healthy volunteers in the UK and 15 healthy volunteers in The Gambia, with no serious adverse events. We have designed our Phase I studies to allow for a vaccination of volunteer groups sequentially with a step-wise increase in mycobacterial exposure, in order to minimize the possibility of a Koch reaction. A Koch reaction describes the development of immunopathology in a person or animal with tuberculosis, when an exaggerated immune response to M.tb is stimulated. It was described in patients with TB disease when Koch performed his original studies employing mycobacteria as a type of therapeutic vaccination. It has now been demonstrated in the mouse model of therapeutic vaccination (Taylor, 2003). Available animal data suggest that these reactions do not occur in mice latently infected with M.tb, suggesting that such reactions may correlate with high bacterial load and that the Koch phenomenon may not pose a problem for vaccination of healthy albeit latently infected humans. We started these studies in healthy volunteers who were as mycobacterially naïve as possible. They were skin test negative and Elispot negative for PPD, ESAT 6 and CFP10, and had not had previously been vaccinated with BCG. We have now completed studies in the UK vaccinating volunteers previously vaccinated with BCG (McShane, submitted). These volunteers are excluded if their Heaf test is greater than grade II. These studies are ongoing in The Gambia. The next group we then plan to vaccinate on this increasing mycobacterial spectrum are healthy volunteers who are latently infected with M.tb. Rationale This study is designed to evaluate the safety of MVA85A in healthy volunteers in the UK who are latently infected with M.tb. A single vaccination with MVA85A, when administered at a dose of 5 x 107pfu intradermally, is safe in both mycobacterially naïve individuals and those previously vaccinated with BCG. We will use the same vaccination regime in this study. Subjects will be defined as being latently infected if they have a positive elispot response to ESAT6 or CFP10. Subjects will be identified from TB contact clinics.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults aged 18 to 50 years
* Resident in or near Oxford for the duration of the vaccination study
* Willingness to allow the investigators to discuss the volunteer's medical history with the volunteer's GP
* Screening Elispot positive (more than 50 spots/million PBMC) for at least any 1 of the 3 ESAT6 peptide pools or any one of the 3 CFP10 pools ; and screening Elispot positive for PPD.
* Heaf test grade II-IV or positive Mantoux test.
* CXR normal; or abnormal but not clinically significant CXR findings with no evidence of past/present TB infection or disease on the CXR.
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day of vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent
* Willingness to undergo an HIV

Exclusion Criteria

* Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis
* Heaf grade IV
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, ε 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Evidence of cardiovascular disease
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of insulin requiring diabetes mellitus
* Chronic or active neurological disease requiring ongoing specialist supervision

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety of a single intradermal injection of 5 x 107pfu MVA85A | One year

SECONDARY OUTCOMES:
Efficacy | One year
latently infected with MVA85A on the immune response, both to antigen 85A (the antigen in
the vaccine) and to ESAT6/CFP10 antigens (M.tb specific).
Endpoints:
The specific endpoints for safety and reactogenicity will be actively and passively collected
data on adverse events (AEs). The specific endpoints for immunogenicity will be markers of
cell-mediated immunity as described below.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839
- [Background] Goonetilleke NP, McShane H, Hannan CM, Anderson RJ, Brookes RH, Hill AV. Enhanced immunogenicity and protective efficacy against Mycobacterium tuberculosis of bacille Calmette-Guerin vaccine using mucosal administration and boosting with a recombinant modified vaccinia virus Ankara. J Immunol. 2003 Aug 1;171(3):1602-9. doi: 10.4049/jimmunol.171.3.1602. PMID 12874255
- [Background] Bejon P, Peshu N, Gilbert SC, Lowe BS, Molyneux CS, Forsdyke J, Lang T, Hill AV, Marsh K. Safety profile of the viral vectors of attenuated fowlpox strain FP9 and modified vaccinia virus Ankara recombinant for either of 2 preerythrocytic malaria antigens, ME-TRAP or the circumsporozoite protein, in children and adults in Kenya. Clin Infect Dis. 2006 Apr 15;42(8):1102-10. doi: 10.1086/501459. Epub 2006 Mar 14. PMID 16575727
- [Background] Huygen K, Content J, Denis O, Montgomery DL, Yawman AM, Deck RR, DeWitt CM, Orme IM, Baldwin S, D'Souza C, Drowart A, Lozes E, Vandenbussche P, Van Vooren JP, Liu MA, Ulmer JB. Immunogenicity and protective efficacy of a tuberculosis DNA vaccine. Nat Med. 1996 Aug;2(8):893-8. doi: 10.1038/nm0896-893. PMID 8705859
- [Background] McShane H, Brookes R, Gilbert SC, Hill AV. Enhanced immunogenicity of CD4(+) t-cell responses and protective efficacy of a DNA-modified vaccinia virus Ankara prime-boost vaccination regimen for murine tuberculosis. Infect Immun. 2001 Feb;69(2):681-6. doi: 10.1128/IAI.69.2.681-686.2001. PMID 11159955
- [Background] Colditz GA, Brewer TF, Berkey CS, Wilson ME, Burdick E, Fineberg HV, Mosteller F. Efficacy of BCG vaccine in the prevention of tuberculosis. Meta-analysis of the published literature. JAMA. 1994 Mar 2;271(9):698-702. PMID 8309034
- [Derived] Tanner R, Kakalacheva K, Miller E, Pathan AA, Chalk R, Sander CR, Scriba T, Tameris M, Hawkridge T, Mahomed H, Hussey G, Hanekom W, Checkley A, McShane H, Fletcher HA. Serum indoleamine 2,3-dioxygenase activity is associated with reduced immunogenicity following vaccination with MVA85A. BMC Infect Dis. 2014 Dec 3;14:660. doi: 10.1186/s12879-014-0660-7. PMID 25466778
- [Derived] Sander CR, Pathan AA, Beveridge NE, Poulton I, Minassian A, Alder N, Van Wijgerden J, Hill AV, Gleeson FV, Davies RJ, Pasvol G, McShane H. Safety and immunogenicity of a new tuberculosis vaccine, MVA85A, in Mycobacterium tuberculosis-infected individuals. Am J Respir Crit Care Med. 2009 Apr 15;179(8):724-33. doi: 10.1164/rccm.200809-1486OC. Epub 2009 Jan 16. PMID 19151191